CLINICAL TRIAL: NCT00622427
Title: Ramelteon for Treatment of Adult Patients With ADHD-Related Insomnia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Takeda (Industry)
Responsible Party: Principal Investigator, Rachel Fargason, MD, Associate Professosr, University of Alabama at Birmingham
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: F071204001
Record Dates: First submitted 2008-02-13; First posted 2008-02-25 (Estimated); Results first posted 2013-05-24 (Estimated); Last update posted 2013-05-24 (Estimated); Status verified 2013-04

CONDITIONS: ADHD With Sleep Onset Insomnia
MeSH Terms: interventions — ramelteon

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ramelteon then placebo (Experimental): 8 mg tablets every night for 2 weeks, then a 2 week washout,then crossover to placebo tablets for 2 weeks.
  Interventions: Drug: Ramelteon
- Placebo then Ramelteon (Experimental): placebo tablets for every night for 2 weeks, then a 2 week washout, followed by 8 mg tablets every night for 2 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ramelteon — 8 mg tablets every night for 2 weeks
  Other Names: Rozerem
  Arms: Ramelteon then placebo
Drug: Placebo — placebo tablets for every night for 2 weeks
  Arms: Placebo then Ramelteon

SUMMARY:
Primary: We hypothesize a clinically significant improvement in sleep latency, sleep-onset and total sleep time measures in adults with ADHD when given a trial of Ramelteon compared to placebo. Secondary:We expect that Ramelteon will show statistically significant improvements vs. placebo in measures of daytime sleepiness and with no decrement in daytime functioning, including such specific items as focus and social and occupational functioning.

DETAILED DESCRIPTION:
Method: 8-week, randomized, double-blind, placebo-controlled crossover trial of Ramelteon in adult ADHD subjects who suffer from initial insomnia.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ADHD and insomnia-
* 19-65 years of age
* In good general health
* Negative pregnancy test

Exclusion Criteria:

* Current primary psychiatric diagnosis other than ADHD
* Positive urine drug screen for any sedative hypnotic or drugs of abuse
* Unstable medical condition
* HIV positive
* Seizure disorder
* Known hypersensitivity to Ramelteon

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2008-02; Primary Completion 2010-02 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were screened by medical and psychiatric history after responding to solicitation with advertisements in local newspapers and from existing clinic populations.
Groups:
- Ramelteon Then Placebo (8 mg): QD for 14 days prior to sleep first, 2 week wash out period, then placebo QD for 14 days prior to sleep
- Placebo Then Ramelteon (8 mg): QD for 14 days prior to sleep first, 2 week wash out period, then Ramelteon QD for 14 days prior to sleep
Period: Overall Study
Arm/Group | Ramelteon Then Placebo (8 mg) | Placebo Then Ramelteon (8 mg)
Started | 16 | 16
Completed | 16 (each subject received 2 weeks of Ramelteon, then 2 weeks of placebo after a two week wash out period) | 16 (each subject received 2 weeks of placebo, then 2 weeks of Ramelteon after a two week wash out period)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ramelteon Then Placebo (8 mg) | Placebo Then Ramelteon (8 mg) | Total
Number analyzed (Participants) | 16 | 16 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 16 | 32
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 6 | 15
  Male | 7 | 10 | 17
Region of Enrollment [Number; unit: participants]
  United States | 16 | 16 | 32

OUTCOME MEASURES:

1. Primary Outcome: Change in Baseline to 2 Weeks ADHD Rating Scale
Description: It is an 18 item scale with 9 symptoms of inattention and 9 symptoms of Impulsivity and Hyperactivity. This scale is the gold standard in assessment of ADHD. Scores range from 0-54. There must be a score of 6 or more in either category to be diagnosed with ADHD. Severity ranges: 6-18 mild, 19-36 moderate, 37-54 severe. The outcome measure is the percentage difference between the total day 1 score for all subjects and the total 14 day score for all subjects.
Time Frame: day 1 to day 14 of study drug
Measure: Mean (Standard Deviation); unit: percentage of change
Groups:
- Ramelteon; Placebo: QD for 14 days prior to sleep first
Arm/Group | Ramelteon | Placebo
Number analyzed (Participants) | 32 | 32
percentage of change | 0 (0) | 0 (0)

2. Secondary Outcome: Change in Clinical Global Impression (CGI)
Description: The CGI is rated on a 7-point scale, with the severity of illness scale using a range of responses from 1 (normal) through to 7 (amongst the most severely ill patients). The outcome measure is the percent difference between the total score for all subjects at day 1 and the total score for all subjects at day 14 of the study drug.
Time Frame: day 1 to day 14 of study drug
Measure: Mean (Standard Deviation); unit: percentage of change
Groups:
- Ramelteon; Placebo: QD for 14 days prior to sleep
Arm/Group | Ramelteon | Placebo
Number analyzed (Participants) | 32 | 32
percentage of change | 0 (0) | 0 (0)

ADVERSE EVENTS:
Time Frame: Length of study--average of 6 weeks
Arm/Group | Ramelteon Then Placebo (8 mg) | Placebo Then Ramelteon (8 mg)
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 3/16 | 4/16
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ramelteon Then Placebo (8 mg) (N=16) | Placebo Then Ramelteon (8 mg) (N=16)
Drowsiness (Nervous system disorders) | 2 (2) | 3 (3)
Hives (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No